CLINICAL TRIAL: NCT07381842
Title: An Investigation of the Effects of Manual Therapy on the Spatiotemporal Gait Characteristics in Patients With Chronic Obstructive Pulmonary Disease
Brief Title: The Effects of Manual Therapy on the Spatiotemporal Gait Characteristics in Patients With Chronic Obstructive Pulmonary Disease
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Aynur Demirel, PT, PhD, Assoc. Prof., Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FTREK25/173
Record Dates: First submitted 2026-01-13; First posted 2026-02-02 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: COPD (Chronic Obstructive Pulmonary Disease); Manuel Therapy; Gait Biomechanics; Muscle Energy Technique; Functional Capacity
Keywords: COPD; Gait; Manuel therapy
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: Participants will be randomized into two group using a computer-based method, taking potential stratification criteria (such as sex, age, and disease severity) into account.
  The Manual Therapy Group and Control Group. After randomization, manual techniques will be applied in patients with COPD in intervention group.
  Study design: Double-blind randomized controlled trial
Who Masked: Participant, Outcomes Assessor
Masking Description: The all participants will be blinded. The outcome assessor who will participate in the gait analysis, balance assessment, and EMG analysis will blind to participant allocation. Participants will be randomized into the intervention and control groups using a computer-based randomization sequence with a 1:1 allocation ratio. Allocation concealment will be ensured using sequentially numbered, sealed, and opaque envelopes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Manual therapy Group (Experimental): Muscle energy techniques and diaphragmatic relaxation techniques
  Interventions: Other: Manual therapy Group
- Control Group (Other): Respiratory exercises and stretching exercises Stretching will be applied to the following muscle groups: pectoralis major and minor, upper trapezius, scalene muscles, sternocleidomastoid, and latissimus dorsi.
  Interventions: Other: Control group

INTERVENTIONS:
Other: Manual therapy Group — For muscle energy techniques, the post-isometric relaxation (PIR) technique will be applied. Participants will be instructed to perform an isometric contraction against mild resistance (20-30% of maximal effort), which will be maintained for 7-10 seconds, followed by a 3-second relaxation period. PIR applications will be performed bilaterally for each muscle group, in 2 sets with a total of 10 repetitions. The muscle groups to which MET will be applied include the pectoralis major and minor, upper trapezius, scalene muscles, sternocleidomastoid, and latissimus dorsi. For the diaphragmatic relaxation technique, the therapist will follow the elevation of the ribs and gently draw the contact points cranially and slightly laterally. During expiration, the therapist will maintain resistance by deepening the contact toward the internal costal margin. The maneuver will be applied in two sets of 10 deep breaths, with a 1-minute rest interval between sets.
  Arms: Manual therapy Group
Other: Control group — Self-stretching and breathing exercise
  Arms: Control Group

SUMMARY:
The primary aim of this study is to investigate the effects of manual therapy on spatiotemporal characteristics of gait and gait variability, functional exercise capacity, and pulmonary function in patients with chronic obstructive pulmonary disease (COPD).

The secondary aims of the study are to determine the effects of manual therapy on balance, respiratory muscle strength, quality of life, physical activity, symptom severity, accessory respiratory muscle activation, peripheral muscle strength, chest wall mobility, dysfunctional breathing, pain, and posture.

DETAILED DESCRIPTION:
Musculoskeletal changes secondary to systemic inflammation in chronic obstructive pulmonary disease (COPD) negatively affect both ventilatory efficiency and ventilation-perfusion matching during walking, leading to a reduction in functional capacity. Current and conventional pulmonary rehabilitation approaches generally aim to improve aerobic capacity, muscle strength, and respiratory muscle endurance. However, aspects such as thoracic spine mobility, costotransverse and costovertebral joint biomechanics, the craniocaudal positioning of the diaphragm, and accessory respiratory muscle activation are still not adequately addressed in existing rehabilitation programs. The effects of manual therapy applied to the thoracic region, trunk, and accessory respiratory muscles on both exercise capacity and the spatiotemporal characteristics of gait have not yet been clearly established. Given the multisystem involvement in COPD, the application of manual therapy-an intervention with a high level of evidence in the management of other musculoskeletal conditions-offers an innovative approach to treatment. It is plausible that muscle energy techniques, one of the manual therapy methods, may reduce hypertonicity in excessively activated accessory respiratory muscles during breathing and thereby enhance chest wall expansion. In the existing literature, the limited number of studies investigating manual therapy interventions in COPD have primarily focused on pulmonary function and exercise capacity; however, there is still no consensus regarding the outcomes. Considering the biomechanical connection between the thoracic cage and the trunk and extremities, it can be hypothesized that manual therapies in COPD may influence gait by affecting lower extremity movements. In this context, manual therapy may impact not only respiratory parameters but also gait performance through the interaction between biomechanics, respiration, and posture in patients with COPD.

ELIGIBILITY:
Inclusion Criteria:

* Age 40 years or older
* Clinically stable for at least the past 4 weeks
* Classified as GOLD stage 1, 2, or 3 according to the Global Initiative for Chronic Obstructive Pulmonary Disease (GOLD) airflow limitation classification
* Classified as group A, B, or E according to the GOLD ABE assessment tool

Exclusion Criteria:

* Use of walking assistive devices
* Receiving long-term oxygen therapy
* Presence of additional orthopedic, neuromuscular, neurological, or cardiac conditions that may affect gait and balance
* History of lung cancer, sarcoidosis, tuberculosis, and/or lung surgery
* Presence of musculoskeletal conditions such as fibromyalgia, rheumatoid arthritis, or osteoarthritis
* Presence of a known mental or cognitive impairment

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2026-02-08 (Estimated); Primary Completion 2026-11-08 (Estimated); Study Completion 2028-01-08 (Estimated)

PRIMARY OUTCOMES:
Spatiotemporal Gait Characteristics (Gait Analysis) | At the baseline and after the eight-week intervention
  The spatiotemporal characteristics of gait and gait variability will be assessed using an electronic walkway system (GAITRite, CIR Systems Inc., Franklin, New Jersey, USA). GAITRite is a system with established reliability and validity for gait assessment in individuals with COPD. Data will be collected at the beginning and at the end of a six-minute walking period. Participants will walk at their self-selected pace. Gait data obtained at the beginning and at the end of the six-minute walk will be averaged for data analysis. Data normalization will be performed using participants' leg length (cm), height (cm), or body weight (kg) values.
Spatial Gait Distance Parameters | At the baseline and after the eight-week intervention
  Mean step length, stride length, and step width measured using the GAITRite electronic walkway system. Unit of Measure: meters (m)
Temporal Gait Parameters | At the baseline and after the eight-week intervention
  Mean stance phase duration, swing phase duration, stride time, and step time assessed using GAITRite.
  Unit of Measure: seconds (s)
Gait Speed | At the baseline and after the eight-week intervention
  Mean walking speed measured using the GAITRite system during self-selected pace walking.
  Unit of Measure: meters per second (m/s)
Cadence | At the baseline and after the eight-week intervention
  Mean cadence assessed using GAITRite during the six-minute walk test. Unit of Measure: steps per minute (steps/min)
Gait Symmetry and Asymmetry Indices | At the baseline and after the eight-week intervention
  Right-left gait symmetry and asymmetry indices derived from spatiotemporal gait parameters.
  Unit of Measure: ratio or percentage (%)
Gait Variability Parameters | At the baseline and after the eight-week intervention
  Stride time variability, step time variability, and step width variability calculated from GAITRite data.
  Unit of Measure: coefficient of variation (%)
Functional exercise capacity | At the baseline and after the eight-week intervention
  Functional exercise capacity will be assessed using the Six-Minute Walk Test (6MWT). The test will be conducted in accordance with the criteria of the American Thoracic Society (ATS). Heart rate and peripheral oxygen saturation (SpO₂) will be measured using a pulse oximeter (Nonin Model 2500C, Nonin Medical, Inc., Plymouth, Minnesota, USA), and blood pressure will be measured using a sphygmomanometer (Erka Perfect Aneroid, Berlin, Germany) before the test, at the first minute, and immediately after the test. Leg fatigue, general fatigue, and dyspnea will be assessed using the Modified Borg Scale. At the end of the test, the total distance walked will be recorded in meters. Predicted values based on age, sex, height, and body weight will be used to calculate the percentage of the predicted walking distance achieved by each participant. To evaluate mechanical workload, the 6MWT workload will be calculated by multiplying the six-minute walking distance by the participant's body weight.
Pulmonary Functions | At baseline and after the eight-week intervention
  Pulmonary functions will be assessed using spirometry in accordance with the guidelines published by the American Thoracic Society (ATS) and the European Respiratory Society (ERS). Forced expiratory volume in one second (FEV₁) will be recorded.
  FEV₁ expressed as a percentage of predicted values based on reference equations. Unit of Measure: Percentage (%)
  Based on spirometry results, airflow limitation in COPD will be classified according to the Global Initiative for Chronic Obstructive Pulmonary Disease (GOLD) criteria, with FEV₁/FVC < 0.70 defined for all groups. Classification will be as follows:
  * GOLD 1 (Mild): FEV₁ ≥ 80% of predicted
  * GOLD 2 (Moderate): 50% ≤ FEV₁ < 80% of predicted
  * GOLD 3 (Severe): 30% ≤ FEV₁ < 50% of predicted
  * GOLD 4 (Very severe): FEV₁ < 30% of predicted
Forced Vital Capacity (FVC) | At the baseline and after the eight-week intervention
  Forced vital capacity (FVC) measured by spirometry following ATS/ERS standards. Unit of Measure: Liters (L) an persantage (%)
FEV₁/FVC Ratio | At the baseline and after the eight-week intervention
  The ratio of forced expiratory volume in one second to forced vital capacity (FEV₁/FVC) obtained from spirometry.
  Unit of Measure: Ratio
Peak Expiratory Flow (PEF) | At the baseline and after the eight-week intervention
  Peak expiratory flow assessed by spirometry according to ATS/ERS guidelines. Unit of Measure: Liters per second (L/s) and persentage (%)
Forced Expiratory Flow 25-75% (FEF₂₅-₇₅) | At the baseline and after the eight-week intervention
  Forced expiratory flow between 25% and 75% of forced vital capacity measured using spirometry.
  Unit of Measure: Liters per second (L/s) and persentage

SECONDARY OUTCOMES:
Respiratory muscle strength | At the baseline and after the eight-week intervention
  Respiratory muscle strength will be determined by measuring maximal inspiratory pressure (MIP) and maximal expiratory pressure (MEP) generated at the mouth using a mouth pressure device (Micro MPM; Micro Medical Ltd., Rochester, UK) with individual antibacterial and antiviral disposable filters.
  For MIP measurement, participants will be instructed to perform a maximal expiration; after the application of a nose clip, they will then perform a maximal inspiration for 1-3 seconds. For MEP measurement, participants will be instructed to perform a maximal inspiration; after the application of a nose clip, they will then perform a maximal expiration for 1-3 seconds.
  The tests will be repeated until no further improvement is observed and the difference between the two best values is less than 5%. The highest value will be recorded. Predicted normal values for respiratory muscle strength will be calculated using age- and sex-specific regression equations.
Peripheral muscle strength | At the baseline and after the eight-week intervention
  Peripheral muscle strength will be assessed using handgrip strength and the one-minute sit-to-stand test. Handgrip strength will be measured using a digital hand dynamometer (Baseline BIMS, Fabrication Enterprises Inc., USA).Participants will be instructed to grip the stabilized dynamometer with maximal force. Measurements will be repeated three times, and the highest value will be recorded.
  Participants will be seated freely on a chair with a height of 46 cm, with the hips and knees flexed at 90°, arms crossed over the chest, and feet positioned at hip width. They will then be instructed to stand up and sit down as many times as possible within one minute at their self-selected pace, without altering body posture. The total number of repetitions will be recorded. This repetition count will be expressed as a percentage of predicted reference values adjusted for sex, height, body weight, and age.
Balance assessment | At the baseline and after the eight-week intervention
  Balance and postural sway will be assessed using a three-component force platform (Bertec Model BP 5050; Bertec Corporation, Columbus, Ohio, USA). Participants will be asked to stand barefoot on the force platform for 10 seconds while maintaining a quiet standing position with a stance width equal to their support base. Postural sway will be evaluated under four different conditions: eyes open and eyes closed on both firm and compliant surfaces. Based on the data, a stability score calculated by the device software will also be expressed as a percentage. Stability limits in the anterior, posterior, right, and left directions will be recorded in centimeters and expressed as percentages.
Accessory Muscle activation | At the baseline and after the eight-week intervention
  Surface electromyography will be used to assess accessory respiratory muscle activation using the Trigno™ system (Delsys Inc., Natick, MA, USA). Four channels will be utilized for data acquisition. To minimize signal crosstalk, electrode placement will be determined in accordance with the recommendations of the Surface Electromyography for the Non-Invasive Assessment of Muscles (SENIAM) guidelines. Activation of the most commonly investigated accessory respiratory muscles will be assessed bilaterally at rest. The muscles evaluated will include the sternocleidomastoid, pectoralis major, upper trapezius, and latissimus dorsi. A standardized maximal voluntary contraction (MVC) protocol will be applied for each muscle. EMG values will be normalized to the MVC obtained for the corresponding muscle and expressed as a percentage of MVC (%MVC).
Posture | At the baseline and after the eight-week intervention
  Posture will be assessed observationally using the evaluation system developed by Corbin et al. Postural deviations will be scored as follows: 0 = none, 1 = mild, 2 = moderate, and 3 = severe. Each region will be evaluated and scored individually, as well as cumulatively. Based on the total score, posture will be categorized into five levels: 0-2 points = excellent, 3-4 points = very good, 5-7 points = good, 8-11 points = fair, and ≥12 points = poor. Higher scores represents worsen posture.
Chest wall assessment | At the baseline and after the eight-week intervention
  Chest wall mobility will be assessed by manual measurement of thoracic expansion using tape. For upper thoracic mobility, the measuring tape will be positioned at the level of the sternal manubrium anteriorly and aligned posteriorly with the T2-T3 vertebrae. Measurement at the mid-thoracic level will be taken at the level of the xiphoid process anteriorly and the T6 vertebra posteriorly. For lower thoracic mobility, the tape will be placed at the level of the costal margin anteriorly and aligned posteriorly with the T10 vertebra. At each measurement level, participants will be instructed to perform maximal inspiration and maximal expiration, and the difference between these two measurements will be recorded as the thoracic expansion value. Measurements will be repeated three times at each level, and the mean of the obtained values will be used for analysis.
Dyspnea Level | At the baseline and after the eight-week intervention
  The Modified Medical Research Council Dyspnea Scale (mMRC) and Dyspnea-12 (D-12) will be used. The mMRC is a five-item scale developed based on various activities that provoke dyspnea. It will be used to assess the level of dyspnea in participants. Individuals will be asked to indicate the activity level that causes breathlessness on the scale. Higher mMRC scores indicate worse dyspnea severity.
  The D-12 is a 12-item instrument that evaluates both the physical and emotional dimensions of breathlessness. Each item is scored on a 0-3 scale, with higher scores indicating more severe dyspnea. The Turkish validity and reliability of the questionnaire have been established.
Severity of symptoms | At the baseline and after the eight-week intervention
  COPD Assessment Test (CAT) will be used. The CAT is an eight-item, unidimensional measure of health status impairment in individuals with COPD. The total score ranges from 0 to 40. A cut-off score of 10 has been defined for the CAT. Higher CAT scores indicate worse symptom severity. Participants will be asked to select the option that best reflects their condition for each item.
  Based on the impact of symptoms on daily life activities, total CAT scores are classified into five categories: >30 points indicate a very high level of impact, >20 points indicate a high level of impact, 10-20 points indicate a moderate level of impact, <10 points indicate a low level of impact, and a score of 5 points is considered the upper limit of normal impact in healthy never-smokers.
Severity of disease | At the baseline and after the eight-week intervention
  The GOLD ABE system will be used. A combined assessment system based on symptom evaluation, spirometric classification, and exacerbation risk is recommended for patients with COPD. According to this combined assessment, patients are categorized into groups A, B, and E.
  * Group A: GOLD stage 1 or 2 (mild or moderate airflow limitation), and/or 0-1 exacerbations per year with no hospitalization due to exacerbation; CAT < 10 or mMRC grade 0-1.
  * Group B: GOLD stage 1 or 2 (mild or moderate airflow limitation), and/or 0-1 exacerbations per year with no hospitalization due to exacerbation; CAT ≥ 10 or mMRC ≥ 2.
  * Group E: GOLD stage 3 or 4 (severe or very severe airflow limitation), and/or ≥ 2 exacerbations per year or ≥ 1 exacerbation leading to hospitalization; mMRC 0-4 and CAT 0-40.
Severity of disease and mortality | At the baseline and after the eight-week intervention
  The BODE Index was developed to assess mortality risk in individuals with COPD. This multidimensional index incorporates body mass index (BMI), airway obstruction (FEV₁ % predicted), dyspnea (mMRC score), and exercise capacity assessed by the six-minute walk distance (6MWD).
  BMI is scored as 0 for values > 21 kg/m² and 1 for values ≤ 21 kg/m². Airway obstruction, reflected by FEV₁ (% predicted), is scored as 0 for values ≥ 65%, 1 for 50-64%, 2 for 36-49%, and 3 for values ≤ 35%. Dyspnea severity based on mMRC scores is scored as 0 for grades 0-1, 1 for grade 2, 2 for grade 3, and 3 for grade 4. Finally, exercise capacity assessed by the 6MWD is scored as 0 for distances ≥ 350 m, 1 for 250-349 m, 2 for 150-249 m, and 3 for distances ≤ 149 m.
  The total BODE score will be calculated by summing the scores obtained from each component. As the total BODE index score increases, the severity of COPD worsens, and prognosis and mortality risk deteriorate.
Quality of life (St. George's Respiratory Questionnaire ) | At the baseline and after the eight-week intervention
  Quality of life will be assessed using the St. George's Respiratory Questionnaire (SGRQ). The Turkish validity and reliability of the questionnaire have been established. The SGRQ is a widely used instrument for individuals with chronic respiratory diseases and consists of three domains: symptoms, activities, and social/psychological impacts. The questionnaire includes a total of 50 items, and scores for each domain as well as the total score are calculated on a scale ranging from 0 to 100, where 0 indicates no limitation or symptoms and 100 indicates the worst health status or maximum limitation. As the SGRQ total score increases, health-related quality of life deteriorates.
Physical Activity (International Physical Activity Questionnaire) | At the baseline and after the eight-week intervention
  Individuals' physical activity levels will be assessed using the International Physical Activity Questionnaire-Short Form (IPAQ-SF). its Turkish validity and reliability were established. For an activity to be considered in the assessment, it must be performed for at least 10 minutes at a time. The IPAQ-SF provides information on time spent sitting, walking, engaging in moderate-intensity activities, and engaging in vigorous-intensity activities. A total score is calculated as MET-minutes per week by multiplying the duration (minutes), frequency (days), and MET (metabolic equivalent) value of each activity. According to the scoring system, physical activity level is classified as low if the total score is less than 600 MET-min/week, moderate if it ranges between 600 and 3000 MET-min/week, high if it exceeds 3000 MET-min/week. As the total IPAQ-SF score increases, the individual's physical activity level improves, with higher MET-minutes per week indicating greater physical activity.
Dysfunctional breathing (The Nijmegen Questionnaire) | At the baseline and after the eight-week intervention
  The Nijmegen Questionnaire will be used to assess respiratory dysfunction and related symptoms. The Turkish validity and reliability of the questionnaire were established by Çakmak et al. (2023). The questionnaire includes 15 items covering respiratory dysfunctions and symptoms such as chest pain, feelings of tension, blurred vision, and shortness of breath. Participants will be asked to indicate the frequency that best represents each symptom on a 0-4 scale (0 = never, 4 = very often). A total score will be calculated. In the Nijmegen Questionnaire, higher total scores indicate greater severity and frequency of respiratory dysfunction symptoms, reflecting more pronounced dysfunctional breathing patterns.
Pain Level (Visual Analog Scale) | At the baseline and after the eight-week intervention
  Thoracic pain intensity will be assessed using the Visual Analog Scale (VAS). The VAS separately evaluates pain at rest, during the night, and during activity. According to this scale, pain is rated on a horizontal straight line measuring 0-10 cm, with the patient marking the point that best represents their pain intensity, resulting in a score between 0 and 10. A score of 0 indicates no pain, whereas a score of 10 represents unbearable pain. Pain intensity will be recorded separately for rest, night-time, and activity-related pain.
  In the Visual Analog Scale (VAS), higher scores indicate greater pain intensity. An increase in the VAS score reflects worsening pain severity, with higher values representing more severe and intolerable pain at rest, during the night, or during activity.

CONTACTS AND LOCATIONS:
Overall Officials: Aynur Demirel, Study Chair — Hacettepe University
Locations (1):
- Hacettepe University, Ankara, Samanpazari, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No